CLINICAL TRIAL: NCT05704881
Title: Monitoring of the End-tidal Carbon Dioxide (EtCO2 ) as a Severity Criterion in COPD Exacerbations: a Prospective Observational Study
Brief Title: Monitoring of the End-tidal Carbon Dioxide (EtCO2) as a Severity Criterion in COPD Exacerbations
Acronym: CO2PD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.077; 2022-A02330-43 (Other: French ethics committees CPP Nord Ouest II)
Record Dates: First submitted 2022-12-19; First posted 2023-01-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Exacerbation Copd
Keywords: Chronic Obstructive Pulmonary Disease; Capnography; COPD exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient admitted for acute Exacerbation of Chronic Obstructive Pulmonary Disease: Patient admitted for acute Exacerbation of COPD. The measurement of EtCO2 will be performed at the emergency department
  Interventions: Diagnostic Test: End-Tidal CO2 measurement during COPD exacerbation

INTERVENTIONS:
Diagnostic Test: End-Tidal CO2 measurement during COPD exacerbation — The EtCO2 will be measured at the emergency reception during assessment of vital signs by the nurse with the help of a mask or oxygen glasses measuring EtCO2. The patient will then be treated conventionally according to current international recommendations. The physician in charge of the patient will be blinded to this measurement. The outcome will be the initiation of invasive or non-invasive ventilation (NIV) within the first 24 hours of admission to the emergency department, as indicated by the physician in charge of the patient.

SUMMARY:
Although we know that these numbers are underestimated, Chronic obstructive pulmonary disease (COPD) is a common chronic respiratory disease that affects between 8 and 12% of adults. According to a 2020 WHO report, it is the third most common cause of mortality in developed countries. This disease is punctuated by exacerbations associated with an 8% mortality of hospitalized patients, increased to 24% when the patient is admitted to intensive care unit. Early detection and treatment of these exacerbations appears to be essential to improve patient survival. End-tidal carbon dioxide (EtCO2) is used to assess a patient's respiratory and hemodynamic status. Indeed, EtCO2 is a non-invasive measure that could allow the estimation of arterial carbon dioxide (PaCO2) without performing blood gases, an arterial blood sampling, classically at the radial artery. This study aimed to find an EtCO2 value which at the time of the initial management, would be predictive of a severe COPD exacerbation, as well as PaCO2.

DETAILED DESCRIPTION:
The study will be conducted in the emergency departments of Grenoble and Lyon University Hospitals.

Patients will be recruited by the dispatch nurse at the emergency department reception according to the inclusion and non-inclusion criteria. The EtCO2 will be measured at the emergency reception during assessment of vital signs by the same nurse with the help of a mask or oxygen glasses measuring EtCO2. The patient will then be treated conventionally according to current international recommendations. The physician in charge of the patient will be blinded to this measurement. Once the patient is discharged from the emergency department, the primary and secondary endpoints will be collected by a clinical research associate 24 hours after admission from medical record.

ELIGIBILITY:
Inclusion Criteria:

* All patient presenting to the emergency department with acute dyspnea and with a history of COPD documented or reported by the patient and/or family
* Male or female≥18 years old who did not oppose to participating in the study

Exclusion Criteria:

* Hypotension (SBP < 90 mmHg or MBP < 65 mmHg)
* Patient already included in the study during a previous visit to the emergency department
* Patient already ventilated with invasive or NIV during admission to the emergency department
* COPD exacerbation rejected after medical and additional examinations
* Non-communicative or non-French speaking patients, or with impaired comprehension, or with impaired consciousness
* Protected persons referred to in articles L1121-6 and L1121-8 of French public health code (deprived of liberty, tutorship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to emergency department for acute exacerbation of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Invasive or non-invasive ventilation (NIV) use (hour/min) | 24 hours
  Invasive or non-invasive ventilation (NIV) use (hour/min)

SECONDARY OUTCOMES:
Arterial Blood Gaz measurement | 15 minutes (after emergency admission)
  PaCO2 and pH values
Concordance between EtCO2 (mmHg) and PaCO2 (mmHg) using Bland and Altman graphical method. | 15 minutes (after emergency admission)
  A Bland and Altman graph will be used to estimate the concordance between values of EtCO2 (mmHg) and PaCO2 (mmHg) measured on the first blood gases sample performed in the emergency department.
Concordance between EtCO2 (mmHg) and PvCO2 (mmHg) using Bland and Altman graphical method. | 15 minutes (after emergency admission)
  A Bland and Altman graph will be used to estimate the concordance between values of EtCO2 (mmHg) and PvCO2 (mmHg) measured on the first venous blood sample performed in the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Damien VIGLINO, Prof. MD PhD, Study Director — University Hospital, Grenoble; Nicolas SEGOND, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble, Isère
  - Hospices Civils de Lyon, Lyon, Rhône

IPD SHARING:
Plan to Share IPD: Yes
The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. The minimum anonymized source data for performing the statistical analysis will be made public at the time of publication, with the article, or deposited in an appropriate public database. Other anonymized data may be available from the principal investigator upon reasonable request and with the consent of the sponsor.
  In accordance with the French law n ° 2002-303 of March 4th, 2002, the subjects can be informed, at their request, of the overall results of the research. In this study, the investigators commit to individually communicating the overall results to each subject participating in the research by a short (popularized) summary and associated with a copy of the scientific article.
Supporting Information: Study Protocol, SAP
Time Frame: at the time of publication
Access Criteria: The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. Moreover, In accordance with the French law n ° 2002-303 of March 4th, 2002

REFERENCES:
- [Background] Molinari N, Briand C, Vachier I, Malafaye N, Aubas P, Georgescu V, Roche N, Chanez P, Bourdin A. Hospitalizations for COPD Exacerbations: Trends and Determinants of Death. COPD. 2015;12(6):621-7. doi: 10.3109/15412555.2015.1007931. Epub 2015 Aug 11. PMID 26263032
- [Background] Wang J, Zhang J, Liu Y, Shang H, Peng L, Cui Z. Relationship between end-tidal carbon dioxide and arterial carbon dioxide in critically ill patients on mechanical ventilation: A cross-sectional study. Medicine (Baltimore). 2021 Aug 20;100(33):e26973. doi: 10.1097/MD.0000000000026973. PMID 34414969
- [Background] Kartal M, Goksu E, Eray O, Isik S, Sayrac AV, Yigit OE, Rinnert S. The value of ETCO2 measurement for COPD patients in the emergency department. Eur J Emerg Med. 2011 Feb;18(1):9-12. doi: 10.1097/MEJ.0b013e328337b9b9. PMID 20224417
- [Background] Jabre P, Jacob L, Auger H, Jaulin C, Monribot M, Aurore A, Margenet A, Marty J, Combes X. Capnography monitoring in nonintubated patients with respiratory distress. Am J Emerg Med. 2009 Nov;27(9):1056-9. doi: 10.1016/j.ajem.2008.08.017. PMID 19931750
- [Background] Dogan NO, Sener A, Gunaydin GP, Icme F, Celik GK, Kavakli HS, Temrel TA. The accuracy of mainstream end-tidal carbon dioxide levels to predict the severity of chronic obstructive pulmonary disease exacerbations presented to the ED. Am J Emerg Med. 2014 May;32(5):408-11. doi: 10.1016/j.ajem.2014.01.001. Epub 2014 Jan 15. PMID 24560835
- [Background] Tyagi D, Govindagoudar MB, Jakka S, Chandra S, Chaudhry D. Correlation of PaCO2 and ETCO2 in COPD Patients with Exacerbation on Mechanical Ventilation. Indian J Crit Care Med. 2021 Mar;25(3):305-309. doi: 10.5005/jp-journals-10071-23762. PMID 33790512
- [Background] Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, Williamson PR, Altman DG, Montgomery A, Lim P, Berlin J, Senn S, Day S, Barbachano Y, Loder E. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA. 2017 Dec 19;318(23):2337-2343. doi: 10.1001/jama.2017.18556. PMID 29260229
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Lin LI. A concordance correlation coefficient to evaluate reproducibility. Biometrics. 1989 Mar;45(1):255-68. PMID 2720055
- See also: WHO Top 10 causes of death — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death